CLINICAL TRIAL: NCT05438524
Title: The Performance of MRI Prostate in Men With Different Prostate Health Index (Phi) Values: Can we Save Some MRI Scans?
Brief Title: The Performance of MRI Prostate in Men With Different Prostate Health Index (Phi) Values
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHIU Ka Fung Peter, Associate Professor, Chinese University of Hong Kong
Other Study IDs: CRE 2021.256
Record Dates: First submitted 2022-06-24; First posted 2022-06-30 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to investigate, in a larger cohort of consecutive men, the proportion of abnormal MRI prostate in different phi ranges, and the cancer detected in Chinese men with abnormal MRI. This study aims to evaluate whether MRI prostate can be omitted in men with lower suspicion of prostate cancer.

DETAILED DESCRIPTION:
This is a prospective cohort study recruiting consecutive men with elevated blood test PSA 4-10 ng/mL, normal prostate on digital rectal examination, and result for blood Prostate Health Index (phi) known. A multi-parametric MRI prostate with contrast will be performed in all subjects. MRI prostate will be reported according to PI-RADS (Prostate Imaging-Reporting and Data Systems) v2.1 recommendations[10] and scored from 1 to 5. A PI-RADS score of 3-5 is considered abnormal. The proportion of abnormal MRI in different phi ranges (primary outcome) will be compared.

The subjects will be offered a prostate biopsy according to usual clinical indications in our hospital: In men with phi >35 (higher risk of significant prostate cancer), prostate biopsy (systematic biopsy, plus MRI-guided if abnormal MRI) will be offered. In men with phi < 35 (lower risk of prostate cancer), prostate biopsy (systematic plus MRI-guided) will be offered only if MRI is abnormal.

ELIGIBILITY:
Inclusion Criteria:

* Ethnically Chinese Men ≥18 years of age
* Clinical suspicion of prostate cancer and indicated for prostate biopsy
* Serum Prostate-specific antigen (PSA) 4-10 ng/mL
* Serum Prostate health index (phi) result available
* Normal Digital rectal examination
* Able to provide written informed consent

Exclusion Criteria:

* Past or current history of prostate cancer
* On 5-alpha reductase inhibitor in the past 6 months (e.g. Finasteride, Dutasteride)
* MRI prostate performed in past 5 years
* Contraindicated to undergo MRI scan (e.g. pacemaker in-situ, claustrophobia, estimated glomerular filtration rate < 50ml/min in serum renal function test within 3 months)
* Contraindicated for prostate biopsy (e.g. uncorrectable coagulopathy, active infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men with elevated PSA of 4-10 ng/mL who were referred to the Urology clinic without prior prostate biopsy, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
In men with higher risk of significant prostate cancer, proportion of men with abnormal MRI at different Prostate Health Index (phi) ranges | Baseline (only one-time point)
  In men with higher risk (phi>35) of significant prostate cancer), proportion of men with abnormal MRI.
In men with lower risk of significant prostate cancer, proportion of men with abnormal MRI at different Prostate Health Index (phi) ranges | Baseline (only one-time point)
  In men with lower risk (phi<35) of significant prostate cancer), proportion of men with abnormal MRI.

SECONDARY OUTCOMES:
Sensitivity of various phi cutoffs to predict PI-RADS score ≥3 in MRI prostate | Baseline (only one-time point)
  Assessed by phi values and PI-RADS score in MRI prostate
Sensitivity of various phi cutoffs to predict PI-RADS score ≥4 in MRI prostate | Baseline (only one-time point)
  Assessed by phi values and PI-RADS score in MRI prostate
Proportion of low risk group diagnosis of clinically significant prostate cancer with abnormal MRI | Baseline (only one-time point)
  Diagnosis of clinically significant prostate cancer (Gleason 3+4 or above) in men with abnormal MRI and phi <35

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ka-Fung CHIU, FRCS, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Culp MB, Soerjomataram I, Efstathiou JA, Bray F, Jemal A. Recent Global Patterns in Prostate Cancer Incidence and Mortality Rates. Eur Urol. 2020 Jan;77(1):38-52. doi: 10.1016/j.eururo.2019.08.005. Epub 2019 Sep 5. PMID 31493960
- [Background] Chan SY, Ng CF, Lee KW, Yee CH, Chiu PK, Teoh JY, Hou SS. Differences in cancer characteristics of Chinese patients with prostate cancer who present with different symptoms. Hong Kong Med J. 2017 Feb;23(1):6-12. doi: 10.12809/hkmj164875. Epub 2016 Dec 9. PMID 27932742
- [Background] Wong HF, Yee CH, Teoh JY, Chan SY, Chiu PK, Cheung HY, Hou SS, Ng CF. Time trend and characteristics of prostate cancer diagnosed in Hong Kong (China) in the past two decades. Asian J Androl. 2019 Jan 1;21(1):104-106. doi: 10.4103/aja.aja_75_18. No abstract available. PMID 30178778
- [Background] Presti JC Jr, O'Dowd GJ, Miller MC, Mattu R, Veltri RW. Extended peripheral zone biopsy schemes increase cancer detection rates and minimize variance in prostate specific antigen and age related cancer rates: results of a community multi-practice study. J Urol. 2003 Jan;169(1):125-9. doi: 10.1016/S0022-5347(05)64051-7. PMID 12478119
- [Background] Carter HB, Hamper UM, Sheth S, Sanders RC, Epstein JI, Walsh PC. Evaluation of transrectal ultrasound in the early detection of prostate cancer. J Urol. 1989 Oct;142(4):1008-10. doi: 10.1016/s0022-5347(17)38971-1. PMID 2677409
- [Background] Chiu PK, Alberts AR, Venderbos LDF, Bangma CH, Roobol MJ. Additional benefit of using a risk-based selection for prostate biopsy: an analysis of biopsy complications in the Rotterdam section of the European Randomized Study of Screening for Prostate Cancer. BJU Int. 2017 Sep;120(3):394-400. doi: 10.1111/bju.13913. Epub 2017 Jun 5. PMID 28498624
- [Background] Chiu PK, Ng CF, Semjonow A, Zhu Y, Vincendeau S, Houlgatte A, Lazzeri M, Guazzoni G, Stephan C, Haese A, Bruijne I, Teoh JY, Leung CH, Casale P, Chiang CH, Tan LG, Chiong E, Huang CY, Wu HC, Nieboer D, Ye DW, Bangma CH, Roobol MJ. A Multicentre Evaluation of the Role of the Prostate Health Index (PHI) in Regions with Differing Prevalence of Prostate Cancer: Adjustment of PHI Reference Ranges is Needed for European and Asian Settings. Eur Urol. 2019 Apr;75(4):558-561. doi: 10.1016/j.eururo.2018.10.047. Epub 2018 Nov 2. PMID 30396635
- [Background] Chiu PK, Roobol MJ, Nieboer D, Teoh JY, Yuen SK, Hou SM, Yiu MK, Ng CF. Adaptation and external validation of the European randomised study of screening for prostate cancer risk calculator for the Chinese population. Prostate Cancer Prostatic Dis. 2017 Mar;20(1):99-104. doi: 10.1038/pcan.2016.57. Epub 2016 Nov 29. PMID 27897172
- [Background] Turkbey B, Rosenkrantz AB, Haider MA, Padhani AR, Villeirs G, Macura KJ, Tempany CM, Choyke PL, Cornud F, Margolis DJ, Thoeny HC, Verma S, Barentsz J, Weinreb JC. Prostate Imaging Reporting and Data System Version 2.1: 2019 Update of Prostate Imaging Reporting and Data System Version 2. Eur Urol. 2019 Sep;76(3):340-351. doi: 10.1016/j.eururo.2019.02.033. Epub 2019 Mar 18. PMID 30898406
- [Background] Alberts AR, Roobol MJ, Verbeek JFM, Schoots IG, Chiu PK, Osses DF, Tijsterman JD, Beerlage HP, Mannaerts CK, Schimmoller L, Albers P, Arsov C. Prediction of High-grade Prostate Cancer Following Multiparametric Magnetic Resonance Imaging: Improving the Rotterdam European Randomized Study of Screening for Prostate Cancer Risk Calculators. Eur Urol. 2019 Feb;75(2):310-318. doi: 10.1016/j.eururo.2018.07.031. Epub 2018 Aug 3. PMID 30082150
- [Background] Drost FH, Osses DF, Nieboer D, Steyerberg EW, Bangma CH, Roobol MJ, Schoots IG. Prostate MRI, with or without MRI-targeted biopsy, and systematic biopsy for detecting prostate cancer. Cochrane Database Syst Rev. 2019 Apr 25;4(4):CD012663. doi: 10.1002/14651858.CD012663.pub2. PMID 31022301
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Kasivisvanathan V, Rannikko AS, Borghi M, Panebianco V, Mynderse LA, Vaarala MH, Briganti A, Budaus L, Hellawell G, Hindley RG, Roobol MJ, Eggener S, Ghei M, Villers A, Bladou F, Villeirs GM, Virdi J, Boxler S, Robert G, Singh PB, Venderink W, Hadaschik BA, Ruffion A, Hu JC, Margolis D, Crouzet S, Klotz L, Taneja SS, Pinto P, Gill I, Allen C, Giganti F, Freeman A, Morris S, Punwani S, Williams NR, Brew-Graves C, Deeks J, Takwoingi Y, Emberton M, Moore CM; PRECISION Study Group Collaborators. MRI-Targeted or Standard Biopsy for Prostate-Cancer Diagnosis. N Engl J Med. 2018 May 10;378(19):1767-1777. doi: 10.1056/NEJMoa1801993. Epub 2018 Mar 18. PMID 29552975
- [Background] Chiu PK, Roobol MJ, Teoh JY, Lee WM, Yip SY, Hou SM, Bangma CH, Ng CF. Prostate health index (PHI) and prostate-specific antigen (PSA) predictive models for prostate cancer in the Chinese population and the role of digital rectal examination-estimated prostate volume. Int Urol Nephrol. 2016 Oct;48(10):1631-7. doi: 10.1007/s11255-016-1350-8. Epub 2016 Jun 27. PMID 27349564
- [Background] Kim L, Boxall N, George A, Burling K, Acher P, Aning J, McCracken S, Page T, Gnanapragasam VJ. Clinical utility and cost modelling of the phi test to triage referrals into image-based diagnostic services for suspected prostate cancer: the PRIM (Phi to RefIne Mri) study. BMC Med. 2020 Apr 17;18(1):95. doi: 10.1186/s12916-020-01548-3. PMID 32299423
- [Background] Epstein JI, Egevad L, Amin MB, Delahunt B, Srigley JR, Humphrey PA; Grading Committee. The 2014 International Society of Urological Pathology (ISUP) Consensus Conference on Gleason Grading of Prostatic Carcinoma: Definition of Grading Patterns and Proposal for a New Grading System. Am J Surg Pathol. 2016 Feb;40(2):244-52. doi: 10.1097/PAS.0000000000000530. PMID 26492179
- [Background] Chiu PK, Teoh JY, Lee WM, Yee CH, Chan ES, Hou SM, Ng CF. Extended use of Prostate Health Index and percentage of [-2]pro-prostate-specific antigen in Chinese men with prostate specific antigen 10-20 ng/mL and normal digital rectal examination. Investig Clin Urol. 2016 Sep;57(5):336-42. doi: 10.4111/icu.2016.57.5.336. Epub 2016 Aug 31. PMID 27617315
- [Background] Chiu PK, Teoh JY, Chan SY, Chu PS, Man CW, Hou SM, Ng CF. Role of PSA density in diagnosis of prostate cancer in obese men. Int Urol Nephrol. 2014 Dec;46(12):2251-4. doi: 10.1007/s11255-014-0826-7. Epub 2014 Sep 9. PMID 25201460
- See also: Hong Kong Cancer Statistics — http://www3.ha.org.hk/cancereg/pdf/factsheet/2017/prostate_.pdf